CLINICAL TRIAL: NCT00553358
Title: Neo ALTTO (Neoadjuvant Lapatinib and/or Trastuzumab Treatment Optimisation) Study: A Randomised, Multicenter Open-label Phase III Study of Neoadjuvant Lapatinib, Trastuzumab and Their Combination Plus Paclitaxel in Women With HER2/ErbB2 Positive Primary Breast Cancer
Brief Title: Neo ALTTO (Neoadjuvant Lapatinib and/or Trastuzumab Treatment Optimisation) Study
Acronym: Neo ALTTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Breast International Group (Other); SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EGF106903; 2006-000564-81 (EudraCT Number); CLAP016B2302 (Other: Novartis)
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms, Breast
Keywords: Lapatinib; ErbB2+; Early Breast Cancer; Neoadjuvant; breast carcinoma; breast cancer; breast lump; HER2 positive metastatic breast cancer; breast cancer positive for human epidermal growth factor receptor 2 (HER2) HER2 positive metastatic breast cancer; breast cancer progression; estrogen-receptor (ER) positive(+) breast cancer; Paget's disease
MeSH Terms: conditions — Breast Neoplasms; Osteitis Deformans | interventions — Lapatinib; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 Lapatinib (Experimental): 1500 mg lapatinib for 6 weeks followed by lapatinib plus weekly paclitaxel for an additional 12 weeks. After definitive surgery, 3 cycles of adjuvant FEC followed by 34 weeks of adjuvant lapatinib.
  Interventions: Drug: Lapatinib; Drug: Paclitaxel
- Arm 2 Trastuzumab (Active Comparator): 4 mg/kg IV loading dose followed by 2 mg/kg IV weekly trastuzumab for 6 weeks followed by 2 mg/kg trastuzumab plus weekly paclitaxel for an additional 12 weeks. After definitive surgery, 3 cycles of adjuvant FEC followed by 34 weeks of adjuvant trastuzumab (8 mg/kg loading dose followed by 6 mg/kg every 3 weeks).
  Interventions: Biological: Trastuzumab; Drug: Paclitaxel
- Arm 3 Lapatinib plus Trastuzumab (Experimental): 1000 mg lapatinib plus 4 mg/kg IV loading dose followed by 2 mg/kg IV weekly trastuzumab for 6 weeks, followed by 750 mg lapatinib plus 2 mg/kg IV weekly trastuzumab plus weekly paclitaxel for an additional 12 weeks. After definitive surgery, 3 cycles of adjuvant FEC followed by 34 weeks of adjuvant lapatinib (1000 mg) in combination with trastuzumab (8 mg/kg loading dose followed by 6 mg/kg every 3 weeks).
  Interventions: Drug: Lapatinib; Biological: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Lapatinib — Small molecule receptor tyrosine kinase inhibitor
  Arms: Arm 1 Lapatinib; Arm 3 Lapatinib plus Trastuzumab
Biological: Trastuzumab — Therapeutic Monoclonal Antibody
  Arms: Arm 2 Trastuzumab; Arm 3 Lapatinib plus Trastuzumab
Drug: Paclitaxel — antimicrotubule agent

SUMMARY:
This is a randomised, open label multicenter Phase III study comparing the efficacy of neoadjuvant lapatinib plus paclitaxel, versus trastuzumab plus paclitaxel, versus concomitant lapatinib and trastuzumab plus paclitaxel given as neoadjuvant treatment in HER2/ErbB2 over-expressing and/or amplified primary breast cancer.

Patients will be randomised to receive either: lapatinib 1500 mg daily, trastuzumab 4 mg/kg intravenous (IV) load followed by 2 mg/kg IV weekly, or lapatinib 1000 mg daily with trastuzumab 4 mg/kg IV load followed by 2 mg/kg IV weekly for a total of 6 weeks. After this biological window, patients on monotherapy arms will continue on the same targeted therapy plus weekly paclitaxel 80 mg/m^2 for a further 12 weeks, up to definitive surgery. In the combination arm, patients will receive lapatinib 750 mg daily in combination with trastuzumab 2 mg/kg IV plus weekly paclitaxel 80mg/m^2 IV for a further 12 weeks, up to definitive surgery. After surgery, patients will receive three courses of adjuvant chemotherapy with 5-Fluorouracil Epirubicin Cyclophosphamide (FEC) followed by the same targeted therapy as in the biological window of the neoadjuvant setting for a further 34 weeks (in the combination arm, lapatinib dose will be 1000 mg daily in combination with trastuzumab). The planned total duration of the anti-HER2 therapy one year.

Primary objective is to evaluate and compare the rate of pathological complete response (pCR) at the time of surgery in patients with HER2/ErbB2 overexpressing or amplified operable breast cancer randomised to lapatinib followed by lapatinib plus paclitaxel versus trastuzumab followed by trastuzumab plus paclitaxel versus lapatinib in combination with trastuzumab followed by lapatinib, trastuzumab plus paclitaxel.

DETAILED DESCRIPTION:
This was a parallel group, three-arm, randomized, multicenter, open-label phase III study. The study compared the efficacy and tolerability of neoadjuvant lapatinib and paclitaxel, versus trastuzumab and paclitaxel, versus the combination of lapatinib with trastuzumab and paclitaxel given as neoadjuvant treatment in HER2/ErbB2 over-expressing and/or amplified primary breast cancer. Subjects were randomized to receive lapatinib, trastuzumab or lapatinib plus trastuzumab for a total of 6 weeks. After this biological window, subjects continued on the same targeted therapy plus weekly paclitaxel for a further 12 weeks, until definitive surgery (total neoadjuvant therapy duration of 18 weeks). Paclitaxel could be initiated at Week 4 if there is evidence of progressive disease (PD) at that time. Within 6 weeks after surgery, subjects received 3 cycles of adjuvant 5-flourouracil, epirubicin and cyclophosphamide (FEC) followed by the same targeted therapy as in the biological window of the neoadjuvant phase for a further 34 weeks (to complete 52 weeks of anti-HER2 therapy).

After completing 52 weeks of (neo-)/adjuvant anti-HER2 therapy, subjects were scheduled to attend post-treatment follow-up every 3 months during the first year (months 12, 15, 18, 21, and 24), every 6months in Years 3 to 5 inclusive, and annually thereafter up to Year 10. Each subject was to be followed for 10 Years. All subjects were to be followed for EFS and OS up to 10 years from last subject randomized.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Age ≥18 years;
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive breast cancer:
* Primary tumour greater than 2 cm diameter, measured by clinical examination and mammography or echography,
* Any N,
* No evidence of metastasis (M0) (isolated supraclavicular node involvement allowed);
* Over expression and/or amplification of HER2 in the invasive component of the primary tumour [Wolff et al 2006] and confirmed by a certified laboratory prior to randomisation
* Known hormone receptor status.
* Haematopoietic status:
* Absolute neutrophil count ≥ 1,5 x 10^9/L,
* Platelet count ≥ 100 x 10^9/L,
* Hemoglobin at least 9 g/dl,
* Hepatic status:
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (< 2 x ULN) is allowed,
* Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times ULN,
* Alkaline phosphatase ≤ 2.5 times ULN,
* Renal status:
* Creatinine ≤ 2.0 mg/dL,
* Cardiovascular:
* Baseline left ventricular ejection fraction (LVEF) ³ 50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan,
* Negative serum pregnancy test, within 2-weeks (preferably 7 days) prior to randomization (For women of childbearing potential)
* Fertile patients must use effective contraception (barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed)
* Signed informed consent form (ICF)
* Patient accepts to make available tumour samples for submission to central laboratory to conduct translational studies as part of this protocol

Exclusion Criteria:

* Received any prior treatment for primary invasive breast cancer;
* Previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated:
* Basal and squamous cell carcinoma of the skin;
* Carcinoma in situ of the cervix.
* Patients with a prior malignancy diagnosed more than 10 years prior to randomisation may enter the study. Patients must have been curatively treated with surgery alone. Radiation therapy or systemic therapy (chemotherapy or endocrine) are NOT permitted. Prior diagnoses of breast cancer or melanoma are excluded.
* Diagnosis of inflammatory breast cancer;
* Bilateral cancer;
* This criterion has been deleted from the protocol Version 1. Patients with multi-focal cancer are no longer excluded.
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnoea at rest, or chronic therapy with oxygen;
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety;
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug;
* Active or uncontrolled infection;
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded;
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies);
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab or lapatinib or their excipients;
* Pregnant or lactating women;
* Concomitant use of CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2008-01-05 (Actual); Primary Completion 2010-05-27 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (102):
- Argentina (6):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Quilmes
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
- Brazil (3):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
- France (9):
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Levallois-Perret
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (17):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Fürstenwalde, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Celle, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Stralsund, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Witten, North Rhine-Westphalia
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Wan Chai
- Novartis Investigative Site, Budapest, Hungary
- India (6):
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Pune
- Italy (7):
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Lecco, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Monza, Lombardy
  - Novartis Investigative Site, Sondrio, Lombardy
  - Novartis Investigative Site, Trento, Trentino-Alto Adige
- Novartis Investigative Site, Vilnius, Lithuania
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Karachi, Pakistan
- Novartis Investigative Site, Lima, Peru
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
- South Africa (4):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Athlone Park, Amanzimtoti
  - Novartis Investigative Site, Capital Park
  - Novartis Investigative Site, Parktown
- South Korea (2):
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Songpa-gu, Seoul
- Spain (10):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Mataró
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Toledo
  - Novartis Investigative Site, Torrevieja (Alicante)
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Gothenburg, Sweden
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Ukraine (9):
  - Novartis Investigative Site, Chernivtsi
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kiev
  - Novartis Investigative Site, Kryvyi Rih
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Simferopol
- United Kingdom (4):
  - Novartis Investigative Site, Epping, Essex
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Background] Baselga J, Piccart M, Gelber R, di CosimoS, Viale G, Koehler M, Rojo F. Neo-ALTTO (Neoadjuvant Lapatinib and/or Trastuzumab Treatment Optimisation) study [BIG 1-06 /solti/EGF106903]: a phase III translational study for HER2-overexpressing early breast cancer. [Lancet]. 2012;S140-6736(11):
- [Derived] Rediti M, Venet D, Joaquin Garcia A, Maetens M, Vincent D, Majjaj S, El-Abed S, Di Cosimo S, Ueno T, Izquierdo M, Piccart M, Pusztai L, Loi S, Salgado R, Viale G, Rothe F, Sotiriou C. Identification of HER2-positive breast cancer molecular subtypes with potential clinical implications in the ALTTO clinical trial. Nat Commun. 2024 Nov 29;15(1):10402. doi: 10.1038/s41467-024-54621-3. PMID 39613746
- [Derived] Chumsri S, Li Z, Serie DJ, Norton N, Mashadi-Hossein A, Tenner K, Brauer HA, Warren S, Danaher P, Colon-Otero G, Partridge AH, Carey LA, Hilbers F, Van Dooren V, Holmes E, Di Cosimo S, Werner O, Huober JB, Dueck AC, Sotiriou C, Saura C, Moreno-Aspitia A, Knutson KL, Perez EA, Thompson EA. Adaptive immune signature in HER2-positive breast cancer in NCCTG (Alliance) N9831 and NeoALTTO trials. NPJ Breast Cancer. 2022 May 24;8(1):68. doi: 10.1038/s41523-022-00430-0. PMID 35610260
- [Derived] Pizzamiglio S, Cosentino G, Ciniselli CM, De Cecco L, Cataldo A, Plantamura I, Triulzi T, El-Abed S, Wang Y, Bajji M, Nuciforo P, Huober J, Ellard SL, Rimm DL, Gombos A, Daidone MG, Verderio P, Tagliabue E, Di Cosimo S, Iorio MV. What if the future of HER2-positive breast cancer patients was written in miRNAs? An exploratory analysis from NeoALTTO study. Cancer Med. 2022 Jan;11(2):332-339. doi: 10.1002/cam4.4449. Epub 2021 Dec 17. PMID 34921525
- [Derived] Powles RL, Redmond D, Sotiriou C, Loi S, Fumagalli D, Nuciforo P, Harbeck N, de Azambuja E, Sarp S, Di Cosimo S, Huober J, Baselga J, Piccart-Gebhart M, Elemento O, Pusztai L, Hatzis C. Association of T-Cell Receptor Repertoire Use With Response to Combined Trastuzumab-Lapatinib Treatment of HER2-Positive Breast Cancer: Secondary Analysis of the NeoALTTO Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):e181564. doi: 10.1001/jamaoncol.2018.1564. Epub 2018 Nov 8. PMID 29902299
- [Derived] Fumagalli D, Venet D, Ignatiadis M, Azim HA Jr, Maetens M, Rothe F, Salgado R, Bradbury I, Pusztai L, Harbeck N, Gomez H, Chang TW, Coccia-Portugal MA, Di Cosimo S, de Azambuja E, de la Pena L, Nuciforo P, Brase JC, Huober J, Baselga J, Piccart M, Loi S, Sotiriou C. RNA Sequencing to Predict Response to Neoadjuvant Anti-HER2 Therapy: A Secondary Analysis of the NeoALTTO Randomized Clinical Trial. JAMA Oncol. 2017 Feb 1;3(2):227-234. doi: 10.1001/jamaoncol.2016.3824. PMID 27684533
- [Derived] Salgado R, Denkert C, Campbell C, Savas P, Nuciforo P, Aura C, de Azambuja E, Eidtmann H, Ellis CE, Baselga J, Piccart-Gebhart MJ, Michiels S, Bradbury I, Sotiriou C, Loi S. Tumor-Infiltrating Lymphocytes and Associations With Pathological Complete Response and Event-Free Survival in HER2-Positive Early-Stage Breast Cancer Treated With Lapatinib and Trastuzumab: A Secondary Analysis of the NeoALTTO Trial. JAMA Oncol. 2015 Jul;1(4):448-54. doi: 10.1001/jamaoncol.2015.0830. PMID 26181252
- [Derived] Nuciforo PG, Aura C, Holmes E, Prudkin L, Jimenez J, Martinez P, Ameels H, de la Pena L, Ellis C, Eidtmann H, Piccart-Gebhart MJ, Scaltriti M, Baselga J. Benefit to neoadjuvant anti-human epidermal growth factor receptor 2 (HER2)-targeted therapies in HER2-positive primary breast cancer is independent of phosphatase and tensin homolog deleted from chromosome 10 (PTEN) status. Ann Oncol. 2015 Jul;26(7):1494-500. doi: 10.1093/annonc/mdv175. Epub 2015 Apr 7. PMID 25851628
- [Derived] de Azambuja E, Holmes AP, Piccart-Gebhart M, Holmes E, Di Cosimo S, Swaby RF, Untch M, Jackisch C, Lang I, Smith I, Boyle F, Xu B, Barrios CH, Perez EA, Azim HA Jr, Kim SB, Kuemmel S, Huang CS, Vuylsteke P, Hsieh RK, Gorbunova V, Eniu A, Dreosti L, Tavartkiladze N, Gelber RD, Eidtmann H, Baselga J. Lapatinib with trastuzumab for HER2-positive early breast cancer (NeoALTTO): survival outcomes of a randomised, open-label, multicentre, phase 3 trial and their association with pathological complete response. Lancet Oncol. 2014 Sep;15(10):1137-46. doi: 10.1016/S1470-2045(14)70320-1. Epub 2014 Aug 14. PMID 25130998
- [Derived] Yarden Y, Pines G. The ERBB network: at last, cancer therapy meets systems biology. Nat Rev Cancer. 2012 Jul 12;12(8):553-63. doi: 10.1038/nrc3309. PMID 22785351
- [Derived] Baselga J, Bradbury I, Eidtmann H, Di Cosimo S, de Azambuja E, Aura C, Gomez H, Dinh P, Fauria K, Van Dooren V, Aktan G, Goldhirsch A, Chang TW, Horvath Z, Coccia-Portugal M, Domont J, Tseng LM, Kunz G, Sohn JH, Semiglazov V, Lerzo G, Palacova M, Probachai V, Pusztai L, Untch M, Gelber RD, Piccart-Gebhart M; NeoALTTO Study Team. Lapatinib with trastuzumab for HER2-positive early breast cancer (NeoALTTO): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2012 Feb 18;379(9816):633-40. doi: 10.1016/S0140-6736(11)61847-3. Epub 2012 Jan 17. PMID 22257673

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg: Oral lapatinib 1000 mg daily plus trastuzumab 4 mg/kg IV load followed by 2 mg/kg IV weekly for 6 weeks, followed by lapatinib 750 mg daily plus trastuzumab (2 mg/kg IV weekly) plus weekly paclitaxel (80 mg/m^2 IV) for an additional 12 weeks
- Lapatinib 1500 mg: Oral lapatinib (1500 milligrams [mg] daily) for 6 weeks, followed by lapatinib plus weekly paclitaxel (80 mg per meters squared [mg/m^2]) intravenous (IV) for an additional 12 weeks
- Trastuzumab 2 mg/kg: Trastuzumab (4 mg/kilograms [kg] IV load followed by 2 mg/kg IV weekly) for 6 weeks, followed by trastuzumab plus weekly paclitaxel (80 mg/m^2 IV) for an additional 12 weeks
Period: Overall Study
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Started | 152 | 154 | 149
Completed (Completed follow-up per protocol event free. Includes subjects who had a follow-up visit or phone call ≥ 9 years + 6 months after randomization and had no EFS events) | 73 | 58 | 61
Not Completed | 79 | 96 | 88
Not completed — Randomized but did not receive treatment | 3 | 3 | 1
Not completed — Lost to Follow-up | 22 | 26 | 18
Not completed — Withdrew completely | 23 | 33 | 34
Not completed — Died during clinical follow-up | 25 | 29 | 32
Not completed — Not dead but were last followed-up prior to 9 years + 6 months after randomization | 4 | 2 | 2
Not completed — Died after clinical follow-up ended | 1 | 2 | 0
Not completed — Withdrew (survival only) - alive at end of survival follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Total
Number analyzed (Participants) | 154 | 149 | 152 | 455
Age, Continuous [Median (Full Range); unit: Years] | 50.0 [28 to 79] | 49.0 [23 to 77] | 50.0 [25 to 80] | 50.0 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 149 | 152 | 455
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 14 | 15 | 42
  Asian - Central/South | 7 | 5 | 5 | 17
  Asian - East | 30 | 28 | 31 | 89
  Asian - South East | 0 | 0 | 2 | 2
  Black or African American/African Heritage | 0 | 4 | 4 | 8
  White - Arabic/North African Heritage | 6 | 5 | 3 | 14
  White - Caucasian European Heritage | 97 | 93 | 92 | 282
  Missing | 1 | 0 | 0 | 1
Number of participants with tumor cells of the indicated histologic grade [Count of Participants; unit: Participants] — Histologic grade, also called differentiation, refers to how much the tumor cells resemble normal cells of the same tissue type.
  Participants
    Well differentiated | 2 | 5 | 5 | 12
    Moderately differentiated | 56 | 53 | 63 | 172
    Poorly differentiated | 73 | 68 | 64 | 205
    Differentiation cannot be assessed | 22 | 23 | 20 | 65
    Missing | 1 | 0 | 0 | 1
Number of participants with lymph nodes (LNs) of the indicated clinical N stage [Count of Participants; unit: Participants] — Clinical N stage is an evaluation/staging of LN status through physical examination. N0, no regional LN metastasis; N1, metastasis to movable ipsilateral axillary LNs (IALNs); N2a, metastasis in IALNs fixed to one another (matted) or the other structures; N2b, metastasis only in clinically apparent ipsilateral internal mammary nodes and in the absence of clinically evident axillary LN metastasis; N3a, metastasis in ipsilateral infraclavicular LNs; N3b, metastasis in ipsilateral internal mammary LNs fixed and axillary LN; N3c, metastasis in ipsilateral subclavicar LNs; Nx, not assessed.
  Participants
    N0 | 34 | 41 | 48 | 123
    N1 | 95 | 85 | 80 | 260
    N2 (including N2a and N2b) | 19 | 13 | 15 | 47
    N3 (including N3a, N3b, and N3c) | 6 | 7 | 6 | 19
    Nx | 0 | 3 | 3 | 6
Number of participants with the indicated IHC results [Count of Participants; unit: Participants] — An Immunohistochemistry (IHC) test gives a score of 0 to 3+, which indicates the amount of Human Epidermal Growth Factor (HER2) receptor proteins on the cancer cells in the sample tissue. A positive score (3+) indicates that HER2 receptor protein is present, a negative score (0-1+) indicates that no HER2 receptor protein is present, and an equivocal score (2+) indicates uncertainty and a result that is open for interpretation. Equivocal results require additional testing. "Not applicable" refers to the number of participants who did not have IHC testing done.
  Participants
    Not applicable | 60 | 53 | 61 | 174
    Equivocal: Score of 2+ | 9 | 5 | 8 | 22
    Positive: Score of 3+ | 81 | 89 | 76 | 246
    Negative: Score of 0-1+ | 0 | 1 | 3 | 4
    Non interpretable | 4 | 1 | 4 | 9
Number of participants with the indicated FISH results [Count of Participants; unit: Participants] — The Fluorescent In Situ Hybridization (FISH) assay was used to determine the overexpression and/or amplification of HER2 in the invasive component of the primary tumor. Amplified indicates that the cell is overexpressing copies of the HER2 gene. Not amplified indicates that there is no overexpression of copies of the HER2 gene. "Not applicable" refers to the number of participants who did not have the FISH assay performed.
  Participants
    Not applicable | 38 | 42 | 41 | 121
    Amplified | 115 | 105 | 109 | 329
    Not amplified | 1 | 2 | 1 | 4
    Not interpretable | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathological Complete Response (pCR) at the Time of Surgery
Description: Pathological complete response is defined as no invasive cancer in the breast or only non-invasive in situ cancer in the breast specimen. Surgical breast and axillary node resection specimens were evaluated for pathologic tumor response according to National Surgical Adjuvant Breast and Bowel Project (NSABP) guidelines, which do not take into account the histological nodal status.
Time Frame: Weeks 20 to 22
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment, except for those who withdrew their consent to use any of their data (permitted by law in certain countries) prior to receiving any study medication
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
participants | 38 | 44 | 78
Statistical Analysis 1: Comparison: Lapatinib 1500 mg vs Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.3416, Binomial; Binomial p-value for Trastuzumab 2 mg/kg versus Lapatinib 1500 mg; Percentage of participants with pCR = -4.85, 97.5% CI 2-sided [-17.6 to 8.16] — Estimation Comments: Estimated value is the difference in the percentage of participants with pCR: Arm1 (Lapatinib 1500 mg) minus Arm2 (Trastuzumab 2 mg/kg)
Statistical Analysis 2: Comparison: Trastuzumab 2 mg/kg vs Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.0001, Binomial; Binomial p-value for Trastuzumab 2 mg/kg versus Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg; Percentage of participants with pCR = 21.79, 97.5% CI 2-sided [9.08 to 34.23] — Estimation Comments: Estimated value is the difference in the percentage of participants with pCR: Arm3 (Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg) minus Arm2 (Trastuzumab 2 mg/kg)

2. Secondary Outcome: Number of Participants With Overall Response at Week 6
Description: The number of participants with overall response (complete response and/or partial response) was evaluated using World Health Organization (WHO) criteria by clinical examination and by mammography and breast echography with bi-dimensional measurements at Week 6. As per WHO criteria: complete response is defined as the disappearance of all lesions; partial response is defined as a greater than 50% decrease in the sum of products of the greatest length and width of the largest lesion; progressive disease is defined as a greater than 25% increase in the sum of products of all measurable lesions.
Time Frame: Week 6
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
participants
  Overall Response | 81 | 45 | 102
  No Change | 57 | 81 | 33
  Progressive Disease | 5 | 11 | 2
  Not Evaluated | 7 | 9 | 12
  Missing Data | 4 | 3 | 3

3. Secondary Outcome: Overall Response at the Time of Surgery
Description: The number of participants with overall response (complete response and/or partial response) was evaluated using WHO criteria by clinical examination and mammography and breast echography with bi-dimensional measurements at the time of surgery (Weeks 20 to 22). As per WHO criteria: complete response is defined as the disappearance of all lesions; partial response is defined as a greater than 50% decrease in the sum of products of the greatest length and width of the largest lesion; progressive disease is defined as a greater than 25% increase in the sum of products of all measurable lesions.
Time Frame: Time of surgery (Weeks 20 to 22)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
participants
  Overall Response | 114 | 105 | 122
  No Change | 8 | 16 | 7
  Progressive Disease | 0 | 2 | 1
  Not Evaluated | 19 | 20 | 14
  Missing Data | 13 | 6 | 8

4. Secondary Outcome: Number of Participants With Negative Lymph Nodes at the Time of Surgery
Description: Participants were assessed for node-negative lymph nodes at the time of surgery. As per the pathological TNM (Tumor, Node, Metastases) classification (pTNM) of malignant tumors: pN, absence or presence and extent of regional lymph node metastasis. Node-negative (pN0) participants had no regional lymph node metastasis. Although not assessed in this measure, pT is the extent of primary tumor, and pM is the absence or presence of distant metastasis.
Time Frame: Time of surgery (Weeks 20 to 22)
Population: ITT Population. Participants with a lymph node status of pNX (i.e., regional lymph nodes cannot be assessed) were omitted from the analysis of node-negative participants.
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 139 | 140 | 137
participants | 72 | 82 | 100

5. Secondary Outcome: Number of Participants With Actual Indicated Surgery
Description: Participants were assessed for the type of surgery they underwent for breast cancer. Non-conservative surgery is defined as a radical or modified radical mastectomy. Conservative surgery is comprised of a lumpectomy, a quadrantectomy/segmentectomy, or a partial mastectomy. Participants who were not assessed as being candidates for non-conservative or conservative surgery were classified as non-operable.
Time Frame: At surgery (Weeks 20 to 22)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
participants
  Conservative | 66 | 58 | 63
  Non-conservative | 77 | 85 | 80
  Non-operable | 11 | 6 | 9

6. Secondary Outcome: Mean Change From Baseline in Tumor Size at Week 6 and at Surgery
Description: Mean change from baseline in tumor in tumor size. Change from baseline in tumor size was defined as tumor size at Week 6/ surgery (Weeks 20 to 22) minus tumor size at baseline. The difference in treatment arms was estimated for Lapatinib 1500 mg versus Trastuzumab 2 mg/kg and for Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg versus Trastuzumab 2 mg/kg.
Time Frame: Week 6 and surgery (Weeks 20 to 22)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
millimeters
  Week 6 | -20.45 (18.43) | -13.42 (16.44) | -25.77 (19.91)
  Surgery (Weeks 20 to 22) | -41.01 (23.81) | -35.47 (22.95) | -43.59 (26.88)

7. Secondary Outcome: Number of Participants Starting Paclitaxel Before Completing 6 Weeks of Treatment With Either Lapatinib or Trastuzumab
Description: Participants with progressive disease at 4 week assessment that were permitted to commence treatment with paclitaxel.
Time Frame: Week 6
Population: ITT Population. Participants who did not start any treatment were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 149 | 146 | 149
participants | 8 | 12 | 6

8. Secondary Outcome: Event-free Survival (EFS) - Median Clinical Follow-up
Description: Event free survival (EFS) is defined as the time from randomization to first EFS event. For subjects who had breast cancer surgery, EFS events were post-surgery breast cancer relapse, second primary malignancy or death without recurrence. For subjects who did not have breast cancer surgery, EFS events were death during clinical follow-up or non-completion of any neoadjuvant investigational product due to disease progression.
Time Frame: From randomization up to approximately year 10
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Number analyzed (Participants) | 152 | 154 | 149
years | 9.69 [9.55 to 9.73] | 9.60 [8.21 to 9.69] | 9.66 [9.50 to 9.72]

9. Secondary Outcome: Event-free Survival (EFS) - Events and Censoring
Description: as for outcome 8
Time Frame: From randomization up to approximately year 10
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Number analyzed (Participants) | 152 | 154 | 149
Number of Participants
  Number of subjects with EFS events | 43 | 47 | 47
  Number of subjects censored - total | 109 | 107 | 102
  Number of subjects censored - Clinical follow-up ongoing | 0 | 0 | 0
  Number of subjects censored - Clinical follow-up ended - total | 103 | 105 | 99
  Number of subjects censored -Clinical follow-up ended - Completed study follow-up | 61 | 49 | 58
  Number of subjects censored - Clinical follow-up ended - Lost to follow-up | 17 | 20 | 10
  Number of subjects censored - Clinical follow-up ended - Withdrew (but consent for survival f/u) | 3 | 6 | 4
  Number of subjects censored - Clinical follow-up ended - Withdrew | 22 | 30 | 27
  Number of subjects censored - Other | 6 | 2 | 3
Statistical Analysis 1: Comparison: Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg vs Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.548, Regression, Cox — The two-sided stratified log-rank test was implemented as the score test from the Cox model; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.57 to 1.34] — Cox models (Cox, 1972), with the stratification factors entered as strata variables, were used to calculate hazard ratios and corresponding confidence intervals for the pairwise comparisons of individual treatment arms with the trastuzumab alone arm
Statistical Analysis 2: Comparison: Lapatinib 1500 mg vs Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.981, Regression, Cox — The two-sided stratified log-rank test was implemented as the score test from the Cox model; Hazard Ratio (HR) = 1.005, 95% CI 2-sided [0.66 to 1.52] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Overall Survival (OS) - Median Survival Follow-up
Description: Overall survival is defined as the period from randomization until death (from any cause). OS was assessed annually for up to 10 years after the randomization of the last participant into the study.
Time Frame: From randomization up to approximately year 10
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Number analyzed (Participants) | 152 | 154 | 149
years | 9.70 [9.60 to 9.76] | 9.62 [8.86 to 9.67] | 9.64 [9.35 to 9.71]

11. Secondary Outcome: Overall Survival (OS) - Deaths and Censoring
Description: as for outcome 10
Time Frame: From randomization up to approximately year 10
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Number analyzed (Participants) | 152 | 154 | 149
Number of Participants
  Number of deaths due to any cause | 26 | 31 | 32
  Number of subjects censored - total | 126 | 123 | 117
  Number of subjects censored - Survival follow-up ongoing | 0 | 0 | 0
  Number of subjects censored - Survival follow-up ended - total | 120 | 121 | 114
  Number of subjects censored -Survival follow-up ended - Completed study follow-up | 74 | 59 | 62
  Number of subjects censored - Survival follow-up ended - Lost to follow-up | 22 | 27 | 18
  Number of subjects censored - Survival follow-up ended - Withdrew | 24 | 35 | 34
  Number of subjects censored - Other | 6 | 2 | 3
Statistical Analysis 1: Comparison: Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg vs Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.379, Regression, Cox — The two-sided stratified log-rank test was implemented as the score test from the Cox model; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.46 to 1.34] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Lapatinib 1500 mg vs Trastuzumab 2 mg/kg; Test type: Superiority or Other; p = 0.880, Regression, Cox — The two-sided stratified log-rank test was implemented as the score test from the Cox model; Hazard Ratio (HR) = 0.962, 95% CI 2-sided [0.58 to 1.60] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Assess Associations Between Locoregional Pathological Complete Response (pCR) and Event-free Survival (EFS) - Median Clinical Follow-up (EFS Landmark Population)
Description: The landmark date is 30 weeks after a subject's randomization. Subjects with missing pCR status were not included in the landmark analysis.
  Clinical follow-up is the period during which the patient is monitored such that all recurrence or second primary malignancy (SPM) or contralateral breast cancer (CBC) events would be reported. Patients are considered in clinical follow-up from randomisation until one of the following occurs: lost to follow-up, withdrawal of consent, end of follow-up due to completion of year 10 visit, termination of study follow-up, or death.
Time Frame: up to year 10
Population: For EFS, the landmark population was the subset of the ITT population who have not had an EFS event within 30 weeks after randomization and were still in clinical follow-up.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Pathological Complete Response (pCR): locoregional pathological Complete Response (pCR)
- No Pathological Complete Response (pCR): no locoregional pathological Complete Response (pCR)
- Overall: Overall - of the 3 arms
Arm/Group | Pathological Complete Response (pCR) | No Pathological Complete Response (pCR) | Overall
Number analyzed (Participants) | 136 | 274 | 410
years
  Median clinical follow-up - all subjects in the EFS landmark analysis | 9.05 [8.86 to 9.14] | 9.11 [9.05 to 9.14] | 9.09 [9.03 to 9.13]
  Median clinical follow-up- EFS landmark analysis - lapatinib + trastuzumab arm (n=67,71,138): number analyzed (Participants) | 67 | 71 | 138
  Median clinical follow-up- EFS landmark analysis - lapatinib + trastuzumab arm (n=67,71,138) | 9.13 [8.97 to 9.23] | 9.10 [7.24 to 9.15] | 9.12 [8.97 to 9.15]
  Median clinical follow-up - subjects in the EFS landmark analysis - lapatinib arm (n=30,104,134): number analyzed (Participants) | 30 | 104 | 134
  Median clinical follow-up - subjects in the EFS landmark analysis - lapatinib arm (n=30,104,134) | 8.08 [6.08 to 9.12] | 9.09 [8.52 to 9.19] | 9.05 [8.23 to 9.12]
  Median clinical follow-up - subjects in the EFS landmark analysis - trastuzumab arm (n=39,99,138): number analyzed (Participants) | 39 | 99 | 138
  Median clinical follow-up - subjects in the EFS landmark analysis - trastuzumab arm (n=39,99,138) | 8.98 [8.38 to 9.21] | 9.12 [9.03 to 9.25] | 9.11 [8.96 to 9.17]
Statistical Analysis 1: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Overall - All subjects in the EFS landmark analysis; Test type: Superiority; p = 0.00079, Regression, Cox; Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.31 to 0.73] — Cox models (Cox, 1972), with the stratification factors entered as strata variables, were used to calculate a hazard ratio and corresponding confidence interval comparing pCR and no pCR
Statistical Analysis 2: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the EFS landmark analysis in the lapatinib + trastuzumab arm; Test type: Superiority; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 0.350, 95% CI 2-sided [0.16 to 0.71] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the EFS landmark analysis in the lapatinib arm; Test type: Superiority; p = 0.134, Regression, Cox; Hazard Ratio (HR) = 0.532, 95% CI 2-sided [0.21 to 1.16] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the EFS landmark analysis in the trastuzumab arm; Test type: Superiority; p = 0.163, Regression, Cox; Hazard Ratio (HR) = 0.601, 95% CI 2-sided [0.28 to 1.20] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Assess Associations Between Locoregional Pathological Complete Response (pCR) and Event-free Survival (EFS) - Number of Participants With EFS Events (EFS Landmark Population)
Description: The landmark date is 30 weeks after a subject's randomization. Subjects with missing pCR status were not included in the landmark analysis.
  For patients who had breast cancer surgery, EFS events are post-surgery breast cancer relapse, second primary malignancy or death without recurrence. For patients who do not undergo breast cancer surgery, EFS events are death during clinical follow-up or non-completion of any neo-adjuvant investigational product due to disease progression or second primary malignancy or contralateral breast cancer.
Time Frame: up to year 10
Population: as for outcome 12
Measure: Number; unit: Number of participants
Arm/Group | Pathological Complete Response (pCR) | No Pathological Complete Response (pCR) | Overall
Number analyzed (Participants) | 136 | 274 | 410
Number of participants
  All subjects in the EFS landmark analysis with EFS events | 29 | 98 | 127
  Subjects in the EFS landmark analysis - lapatinib + trastuzumab arm with EFS events (n=67,71,138): number analyzed (Participants) | 67 | 71 | 138
  Subjects in the EFS landmark analysis - lapatinib + trastuzumab arm with EFS events (n=67,71,138) | 11 | 28 | 39
  Subjects in the EFS landmark analysis in the lapatinib arm with EFS events (n=30,104,134): number analyzed (Participants) | 30 | 104 | 134
  Subjects in the EFS landmark analysis in the lapatinib arm with EFS events (n=30,104,134) | 7 | 36 | 43
  Subjects in the EFS landmark analysis in the trastuzumab arm with EFS events (n=39,99,138): number analyzed (Participants) | 39 | 99 | 138
  Subjects in the EFS landmark analysis in the trastuzumab arm with EFS events (n=39,99,138) | 11 | 34 | 45

14. Secondary Outcome: Assess Associations Between Locoregional Pathological Complete Response (pCR) and and Overall Survival (OS) - Median Clinical Follow-up (OS Landmark Population)
Description: The landmark date is 30 weeks after a subject's randomization. Subjects with missing pCR status were not included in the landmark analysis.
  Patients are considered in survival follow-up from randomisation until one of the following occurs: lost to follow-up, withdrawal of consent, end of follow-up due to completion of year 10 visit, termination of study follow-up, or death. For subjects with no death recorded in the database, time to death is censored.
Time Frame: up to year 10
Population: For OS, the landmark population was the subset of the ITT population who were alive and were followed up for overall survival 30 weeks after randomization.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Pathological Complete Response (pCR) | No Pathological Complete Response (pCR) | Overall
Number analyzed (Participants) | 137 | 283 | 420
years
  Median survival follow-up - All subjects in the OS landmark analysis | 9.10 [8.97 to 9.18] | 9.09 [9.03 to 9.12] | 9.09 [9.04 to 9.13]
  Median survival follow-up - OS landmark analysis in the lapatinib + trastuzumab arm (n=67,72,139): number analyzed (Participants) | 67 | 72 | 139
  Median survival follow-up - OS landmark analysis in the lapatinib + trastuzumab arm (n=67,72,139) | 9.14 [9.05 to 9.24] | 9.09 [7.95 to 9.15] | 9.12 [9.05 to 9.16]
  Median survival follow-up - OS landmark analysis in the lapatinib (n=30,109,139): number analyzed (Participants) | 30 | 109 | 139
  Median survival follow-up - OS landmark analysis in the lapatinib (n=30,109,139) | 8.31 [7.24 to 9.15] | 9.08 [8.95 to 9.14] | 9.07 [8.50 to 9.12]
  Median survival follow-up - OS landmark analysis in the trastuzumab arm (n=40,102,142): number analyzed (Participants) | 40 | 102 | 142
  Median survival follow-up - OS landmark analysis in the trastuzumab arm (n=40,102,142) | 8.98 [8.02 to 9.21] | 9.09 [8.51 to 9.15] | 9.07 [8.86 to 9.14]
Statistical Analysis 1: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Overall - All subjects in the OS landmark analysis; Test type: Superiority; p = 0.00041, Regression, Cox; Hazard Ratio (HR) = 0.366, 95% CI 2-sided [0.20 to 0.63] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the OS landmark analysis in the lapatinib + trastuzumab arm; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.223, 95% CI 2-sided [0.07 to 0.58] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the OS landmark analysis in the lapatinib arm; Test type: Superiority; p = 0.125, Regression, Cox; Hazard Ratio (HR) = 0.433, 95% CI 2-sided [0.12 to 1.17] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Pathological Complete Response (pCR) vs No Pathological Complete Response (pCR); Subjects in the OS landmark analysis in the trastuzumab arm; Test type: Superiority; p = 0.058, Regression, Cox; Hazard Ratio (HR) = 0.414, 95% CI 2-sided [0.15 to 1.00] — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Assess Associations Between Locoregional Pathological Complete Response (pCR) and and Overall Survival (OS) - Number of Participants Who Died (OS Landmark Population)
Description: The landmark date is 30 weeks after a subject's randomization. Subjects with missing pCR status were not included in the landmark analysis. Includes deaths due to any cause.
Time Frame: up to year 10
Population: as for outcome 14
Measure: Number; unit: Number of Participants
Arm/Group | Pathological Complete Response (pCR) | No Pathological Complete Response (pCR) | Overall
Number analyzed (Participants) | 137 | 283 | 420
Number of Participants
  All participants in the OS landmark analysis who died | 15 | 70 | 85
  Participants in the OS landmark analysis in the lapatinib + trastuzumab arm who died (n=67,72,139): number analyzed (Participants) | 67 | 72 | 139
  Participants in the OS landmark analysis in the lapatinib + trastuzumab arm who died (n=67,72,139) | 5 | 19 | 24
  Participants in the OS landmark analysis in the lapatinib arm who died (n=30,109,139): number analyzed (Participants) | 30 | 109 | 139
  Participants in the OS landmark analysis in the lapatinib arm who died (n=30,109,139) | 4 | 26 | 30
  Participants in the OS landmark analysis in the trastuzumab arm who died (n=40,102,142): number analyzed (Participants) | 40 | 102 | 142
  Participants in the OS landmark analysis in the trastuzumab arm who died (n=40,102,142) | 6 | 25 | 31

16. Secondary Outcome: To Assess Safety Via a Comparison of the Three Treatment Arms - to Measure On-treatment Primary Cardiac Endpoints
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 31 weeks.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
Number analyzed (Participants) | 149 | 151 | 148
Participants | 2 [0.16 to 4.76] | 0 [0.00 to 2.41] | 1 [0.02 to 3.71]

17. Secondary Outcome: Metabolic Response Rate Determined by Positron Emission Tomography/Computed Tomography (PET/CT)
Description: Metabolic Response Rate determined by Positron Emission Tomography/Computed Tomography (PET/CT)
Time Frame: Week 2 and Week 6
Population: Translational Data Set. Note that evaluable samples were not available for all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 26 | 26 | 25
Percentage of participants
  Metabolic Response Rate (%) Determined by PET/CT at week 2 | 66.7 | 56.5 | 95.0
  Metabolic Response Rate (%) Determined by PET/CT at week 6 | 60.9 | 43.5 | 78.9

18. Secondary Outcome: Percentage of Participants With the Indicated Biomarker Expression - PIK3CA.
Description: Biomarker levels of phosphatidylinositol 3-kinase (PI3K) catalytic subunit (PIK3CA) were assessed in participants at baseline.
Time Frame: Baseline
Population: Translational Data Set. Note that evaluable samples were not available for all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 124 | 112 | 119
Percentage of participants | 23 | 19 | 25

19. Secondary Outcome: Percentage of Participants With the Indicated Biomarker Expression - PTEN.
Description: Biomarker levels of phosphate and tensin homolog deleted from chromosome 10 (PTEN) were assessed in participants at baseline.
Time Frame: Baseline
Population: Translational Data Set. Note that evaluable samples were not available for all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 123 | 114 | 112
Percentage of participants
  Biomarker: PTEN by Cell Signalling Technology - PTEN Normal (%) | 74 | 70 | 75
  Biomarker: PTEN by Cell Signalling Technology - PTEN Loss (%) | 26 | 30 | 25

20. Secondary Outcome: Ratio (95% CI) of Geometric Means in p95HER2 Expression in HR Positive Patients With pCR vs no pCR
Description: Ratio (95% CI) of geometric means in p95 human epidermal growth factor receptor (p95HER2) expression in hormone-receptor (HR) positive patients with pathological complete response (pCR) vs no pCR
Time Frame: Baseline
Population: Translational Data Set. Note that evaluable samples were not available for all participants.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 97 | 93 | 91
Ratio | 1.0 [0.50 to 1.87] | 1.6 [1.0 to 2.71] | 2.1 [1.2 to 3.7]

21. Secondary Outcome: Percentage of Participants With Circulating Tumor Cells (CTC) in the Bloodstream
Description: Circulating tumor cells (CTCs) are cells that have detached from a primary tumor and circulate in the bloodstream. In the adjuvant phase, after surgery all participants received 3 courses of adjuvant 5-fluorouracil, epirubicin and cyclophosphamide, followed by lapatinib 1500 mg or trastuzumab 2 mg/kg or lapatinib 1000/750 mg plus trastuzumab 2 mg/kg given prior to surgery in the neoadjuvant setting for an additional 34 weeks.
Time Frame: Measurement performed at one or more of the time points: baseline, week 2 or week 18
Population: Translational Data Set. Note that evaluable samples were not available for all participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 19 | 12 | 20
Percentage of Participants | 21 | 17 | 25

22. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, which was approximately 31 weeks. Deaths post treatment survival follow up were collected after the on treatment period, up to 10 years.
Time Frame: on-treatment: up to week 31; post-treatment: up to year 10
Population: Safety population (for on-treatment deaths) and ITT (for total deaths)
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Trastuzumab 2 mg/kg | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg
Number analyzed (Participants) | 154 | 149 | 152
Participants
  Total Deaths | 31 | 32 | 26
  On-Treatment Deaths (n=151,148,149): number analyzed (Participants) | 151 | 148 | 149
  On-Treatment Deaths (n=151,148,149) | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 31 weeks.
Arm/Group | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg | Lapatinib 1500 mg | Trastuzumab 2 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/149 | 2/151 | 0/148
Serious Adverse Events (participants affected / at risk) | 61/149 | 58/151 | 36/148
Other Adverse Events (participants affected / at risk) | 147/149 | 148/151 | 141/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg (N=149) | Lapatinib 1500 mg (N=151) | Trastuzumab 2 mg/kg (N=148)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 2 | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 14 | 13 | 16
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 9 | 9 | 0
DUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 1 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 1 | 2
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 5 | 2 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4 | 4 | 0
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 15 | 23 | 3
APPENDICITIS (Infections and infestations) | 0 | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1 | 0
BREAST CELLULITIS (Infections and infestations) | 1 | 0 | 1
CELLULITIS (Infections and infestations) | 2 | 1 | 2
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 0 | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 1 | 1
MASTITIS (Infections and infestations) | 1 | 2 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 0 | 2
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 3 | 0
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 | 0 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
POISONING (Injury, poisoning and procedural complications) | 0 | 1 | 0
SEROMA (Injury, poisoning and procedural complications) | 1 | 1 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERPHOSPHATASAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
LOBULAR BREAST CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 1 | 0
NEPHRECTASIA (Renal and urinary disorders) | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1000/750 mg + Trastuzumab 2 mg/kg (N=149) | Lapatinib 1500 mg (N=151) | Trastuzumab 2 mg/kg (N=148)
ANAEMIA (Blood and lymphatic system disorders) | 36 | 33 | 27
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 18 | 10
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 | 2 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 47 | 51 | 37
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 2 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 4 | 0 | 2
PALPITATIONS (Cardiac disorders) | 6 | 6 | 3
TACHYCARDIA (Cardiac disorders) | 4 | 2 | 4
EAR PAIN (Ear and labyrinth disorders) | 3 | 1 | 1
TINNITUS (Ear and labyrinth disorders) | 6 | 1 | 3
VERTIGO (Ear and labyrinth disorders) | 11 | 7 | 6
DRY EYE (Eye disorders) | 4 | 1 | 2
LACRIMATION INCREASED (Eye disorders) | 3 | 3 | 1
VISUAL IMPAIRMENT (Eye disorders) | 2 | 2 | 3
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 | 1 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 10 | 8 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 21 | 28 | 13
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 23 | 27 | 16
ANAL INFLAMMATION (Gastrointestinal disorders) | 4 | 2 | 1
CONSTIPATION (Gastrointestinal disorders) | 18 | 15 | 15
DIARRHOEA (Gastrointestinal disorders) | 128 | 123 | 52
DRY MOUTH (Gastrointestinal disorders) | 9 | 5 | 3
DYSPEPSIA (Gastrointestinal disorders) | 17 | 26 | 10
DYSPHAGIA (Gastrointestinal disorders) | 3 | 0 | 3
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 3 | 2 | 2
FLATULENCE (Gastrointestinal disorders) | 3 | 5 | 2
GASTRITIS (Gastrointestinal disorders) | 2 | 8 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 | 2 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 13 | 10 | 10
MOUTH ULCERATION (Gastrointestinal disorders) | 12 | 4 | 1
NAUSEA (Gastrointestinal disorders) | 75 | 81 | 76
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 | 2 | 0
STOMATITIS (Gastrointestinal disorders) | 27 | 18 | 23
TOOTHACHE (Gastrointestinal disorders) | 4 | 1 | 2
VOMITING (Gastrointestinal disorders) | 54 | 57 | 38
ASTHENIA (General disorders) | 39 | 47 | 35
AXILLARY PAIN (General disorders) | 5 | 0 | 3
CHEST DISCOMFORT (General disorders) | 0 | 3 | 6
CHEST PAIN (General disorders) | 5 | 5 | 6
CHILLS (General disorders) | 11 | 3 | 6
FACE OEDEMA (General disorders) | 3 | 5 | 4
FATIGUE (General disorders) | 52 | 45 | 38
FEELING COLD (General disorders) | 0 | 1 | 3
GENERALISED OEDEMA (General disorders) | 1 | 3 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 2 | 2
MUCOSAL DRYNESS (General disorders) | 3 | 2 | 2
MUCOSAL EROSION (General disorders) | 3 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 36 | 34 | 22
OEDEMA (General disorders) | 4 | 0 | 11
OEDEMA PERIPHERAL (General disorders) | 8 | 9 | 13
PAIN (General disorders) | 3 | 6 | 2
PERIPHERAL SWELLING (General disorders) | 4 | 2 | 3
PYREXIA (General disorders) | 34 | 23 | 23
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 21 | 26 | 7
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 55 | 55 | 39
HYPERSENSITIVITY (Immune system disorders) | 6 | 6 | 7
SEASONAL ALLERGY (Immune system disorders) | 3 | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 5 | 3
CONJUNCTIVITIS (Infections and infestations) | 11 | 8 | 5
CYSTITIS (Infections and infestations) | 8 | 6 | 3
HERPES SIMPLEX (Infections and infestations) | 3 | 0 | 2
INFLUENZA (Infections and infestations) | 8 | 8 | 9
LOCALISED INFECTION (Infections and infestations) | 3 | 3 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 1
MASTITIS (Infections and infestations) | 2 | 1 | 3
NAIL INFECTION (Infections and infestations) | 8 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 11 | 12 | 11
ORAL HERPES (Infections and infestations) | 2 | 0 | 3
PARONYCHIA (Infections and infestations) | 17 | 14 | 2
PHARYNGITIS (Infections and infestations) | 4 | 7 | 5
PUSTULE (Infections and infestations) | 3 | 1 | 1
RHINITIS (Infections and infestations) | 6 | 4 | 5
SINUSITIS (Infections and infestations) | 3 | 5 | 2
SKIN INFECTION (Infections and infestations) | 4 | 1 | 2
TONSILLITIS (Infections and infestations) | 0 | 3 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 9 | 14
URINARY TRACT INFECTION (Infections and infestations) | 11 | 14 | 6
VAGINAL INFECTION (Infections and infestations) | 5 | 1 | 2
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 3
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 16 | 11 | 18
SEROMA (Injury, poisoning and procedural complications) | 2 | 0 | 6
THERMAL BURN (Injury, poisoning and procedural complications) | 3 | 0 | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 4 | 4 | 6
EJECTION FRACTION DECREASED (Investigations) | 6 | 2 | 4
GAMMA-GLUTAMYLTRANSFERASE (Investigations) | 3 | 2 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 7 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 3 | 1 | 2
WEIGHT DECREASED (Investigations) | 8 | 10 | 1
WEIGHT INCREASED (Investigations) | 2 | 2 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 35 | 39 | 17
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 5 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 4
HYPERPHOSPHATASAEMIA (Metabolism and nutrition disorders) | 22 | 22 | 12
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 | 26 | 32
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 | 10 | 14
BONE PAIN (Musculoskeletal and connective tissue disorders) | 10 | 12 | 18
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 | 16 | 11
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 31 | 33 | 34
NECK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 5 | 5
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13 | 20 | 13
AGEUSIA (Nervous system disorders) | 4 | 3 | 0
DIZZINESS (Nervous system disorders) | 13 | 13 | 15
DYSGEUSIA (Nervous system disorders) | 6 | 6 | 1
HEADACHE (Nervous system disorders) | 31 | 27 | 26
HYPOAESTHESIA (Nervous system disorders) | 9 | 7 | 12
MEMORY IMPAIRMENT (Nervous system disorders) | 2 | 4 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 19 | 21 | 19
NEUROTOXICITY (Nervous system disorders) | 3 | 6 | 3
PARAESTHESIA (Nervous system disorders) | 24 | 15 | 22
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 13 | 19 | 14
POLYNEUROPATHY (Nervous system disorders) | 5 | 1 | 3
TASTE DISORDER (Nervous system disorders) | 9 | 6 | 1
ANXIETY (Psychiatric disorders) | 7 | 9 | 11
DEPRESSION (Psychiatric disorders) | 7 | 5 | 9
INSOMNIA (Psychiatric disorders) | 34 | 23 | 24
SLEEP DISORDER (Psychiatric disorders) | 5 | 4 | 2
DYSURIA (Renal and urinary disorders) | 11 | 6 | 5
HAEMATURIA (Renal and urinary disorders) | 4 | 0 | 0
AMENORRHOEA (Reproductive system and breast disorders) | 6 | 3 | 1
BREAST DISCHARGE (Reproductive system and breast disorders) | 3 | 0 | 0
BREAST PAIN (Reproductive system and breast disorders) | 6 | 5 | 15
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 | 2 | 3
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 4
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 2 | 2 | 3
VULVOVAGINAL INFLAMMATION (Reproductive system and breast disorders) | 0 | 4 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 2 | 2 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 25 | 17 | 26
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 13
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 6
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 37 | 30 | 22
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 16 | 20 | 15
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 10
ACNE (Skin and subcutaneous tissue disorders) | 22 | 20 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 95 | 90 | 96
DERMATITIS (Skin and subcutaneous tissue disorders) | 13 | 13 | 8
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 14 | 12 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 28 | 29 | 8
ECZEMA (Skin and subcutaneous tissue disorders) | 6 | 4 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 14 | 14 | 15
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 8 | 4 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 36 | 26 | 18
NAIL DYSTROPHY (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
ONYCHALGIA (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 7 | 0 | 2
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 14 | 14 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 24 | 29 | 9
RASH (Skin and subcutaneous tissue disorders) | 67 | 68 | 28
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 4 | 3 | 3
SCAR PAIN (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 13 | 4 | 4
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 6 | 6 | 2
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
FLUSHING (Vascular disorders) | 1 | 3 | 6
HAEMATOMA (Vascular disorders) | 3 | 1 | 1
HOT FLUSH (Vascular disorders) | 22 | 15 | 21
HYPERTENSION (Vascular disorders) | 5 | 5 | 8
HYPOTENSION (Vascular disorders) | 8 | 5 | 2
LYMPHOEDEMA (Vascular disorders) | 3 | 5 | 3
PHLEBITIS (Vascular disorders) | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety